CLINICAL TRIAL: NCT00880100
Title: Efficacy and Safety of Ultrase MT12 in the Control of Steatorrhea in Cystic Fibrosis (CF) and Pancreatic Insufficient (PI) Children Aged 2 to 6 Years Old
Brief Title: Use of Ultrase® MT12 in Young Cystic Fibrosis Children (CF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMT12CF08-01
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Results first posted 2015-02-19 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency
Keywords: Steatorrhea; Malabsorption of fat; Pancreatic enzymes; Abdominal pain; Greasy stools
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Steatorrhea; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrase® MT12 (Experimental)
  Interventions: Drug: Ultrase® MT12

INTERVENTIONS:
Drug: Ultrase® MT12 — Ultrase® MT12 capsules will be given orally daily based on investigator's discretion to a maximum dose of 2,500 lipase units per kilogram (kg) body weight per meal or snack for 19 to 24 days during the treatment phase. Total maximum dose not to exceed 10,000 lipase units/kg/day.

SUMMARY:
Multicenter, explorative, phase IIIb, open-label study to assess the efficacy and safety of Ultrase® MT12, in the control of steatorrhea and clinical signs and symptoms of malabsorption in CF children with pancreatic insufficiency (PI). This study is sponsored by Aptalis Pharma (formerly Axcan).

DETAILED DESCRIPTION:
This is a multicenter, explorative, phase IIIb, open-label study in patients with CF and PI. The study consists of a screening visit (visit 1), followed by a baseline phase of 9 days (plus a 5-day window if necessary) during which the regular pancreatic enzyme will be maintained and 10 stool samples will be collected over 5 days, for baseline evaluation of steatorrhea. Afterward, a treatment phase of 19 days (plus a 5-day window if necessary) with Ultrase® MT12 will follow (the usual pancreatic enzyme will be replaced by Ultrase® MT12). Over the last 5 days of the treatment phase, 10 additional stool samples will be collected, for evaluation of steatorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 2 to 6 years inclusively
* Patients with current diagnosis of CF based on one or more typical clinical features of CF or a sibling with CF or a positive newborn screening and at least either with sweat chloride test greater than or equal to 60 millimoles/liter (mmol/L) by quantitative pilocarpine iontophoresis on two separate occasions or two identifiable CF-causing mutations
* Patients with presence of PI as demonstrated by fecal elastase (FE-1) less than 100 microgram/gram (mcg/g) of stools (performed by ScheBo test) and requiring pancreatic enzyme supplementation
* Patients who are able to eat a high-fat diet calculated at a value between 2g to 4g fat/kg of body weight per day during the whole study and having a current adequate nutritional status based on the body mass index (BMI) greater than or equal to fifth percentile
* Patients receiving current treatment of PI with pancreatic enzymes
* The parent or legal guardian signed informed consent form (ICF) and is mentally able to understand and comply with the study procedures

Exclusion Criteria:

* Patients currently receiving or received an Ultrase® MT product (MT12, MT18, MT20) for PI in the last 30 days
* Patients having known contraindication, sensitivity or hypersensitivity to Ultrase® or to any porcine protein
* Patients with presence of a medical condition known to increase fecal fat loss or that could compromise study results or the study patient safety
* Patients with current diagnosis or history of complete distal intestinal obstruction syndrome (DIOS) in the past 6 months or who had 2 or more episodes of incomplete DIOS in the past year
* Patients with use of any prohibited medication or product at study entry and during the course of the study
* Patients with chronic use of narcotics
* Patients with use of bowel stimulants and/or laxatives more than once a week
* Patients with presence of acute pancreatitis or exacerbation of chronic pancreatic disease
* Patients with presence of an acute infection that needed to be treated with oral or intravenous (IV) broad-spectrum antibiotics
* Patients having history of significant bowel resection; small bowel resection for meconium ileus at birth and appendectomy were accepted. Patients with Presence of dysmotility disorders
* Patients with presence of chronic or severe abdominal pain
* Patients unable to comply with diet requirement
* Patients receiving enteral tube feeding overnight at study entry or who will need to receive enteral tube feeding overnight during the course of the study
* Patients with history of or a current diagnosis of clinically significant portal hypertension
* Patients with presence of poorly controlled diabetes according to the Investigator's clinical judgment
* Patients having any condition or pre-study laboratory abnormality or history of any illness which, in the opinion of the Investigator, might have put the patient at risk, prevented the patient from completing the study, or otherwise affect the outcome of the study
* Patient with use of any investigational drug within 30 days prior to the date of signature of the ICF

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (15):
- United States (15):
  - The Children's Hospital, Aurora, Colorado
  - University of Michigan Health System Cystic Fibrosis Center, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital-Spectrum Health Research Department, Grand Rapids, Michigan
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Rainbow Babies and Children's Hospital - Cystic Fibrosis Center, Cleveland, Ohio
  - Children's Medical Center of Dayton, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Respiratory Diseases of Children and Adolescents, Oklahoma City, Oklahoma
  - Pennsylvania State University and the Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - UW Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment started in April 2009 and was completed in November 2009. Cystic fibrosis (CF) patients with pancreatic insufficiency (PI), aged 2 to 6 years old inclusively, were enrolled from 14 CF centers located in United States of America.
Groups:
- Ultrase® MT12: Patients received usual pancreatic enzymes therapy for 9 to 14 days during baseline phase followed by Ultrase® MT12 capsules orally daily based on investigator's discretion to a maximum dose of 2,500 lipase units per kilogram (kg) body weight per meal or snack for 19 to 24 days during the treatment phase. Total maximum dose was not to exceed 10,000 lipase units/kg/day.
Period: Baseline Phase-Usual Pancreatic Enzymes
Arm/Group | Ultrase® MT12
Started | 49
Completed | 48
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Treatment Phase With Ultrase® MT12
Arm/Group | Ultrase® MT12
Started | 48
Completed | 45
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: Safety population included patients who signed an informed consent form (ICF), completed the baseline phase and started the treatment phase by taking at least one dose of the study treatment.
Groups:
- Ultrase® MT12: Ultrase® MT12 capsules were given orally daily based on investigator's discretion to a maximum dose of 2,500 lipase units per kilogram (kg) body weight per meal or snack for 19 to 24 days during the treatment phase. Total maximum dose was not to exceed 10,000 lipase units/kg/day.
Arm/Group | Ultrase® MT12
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.8 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Control of Steatorrhea
Description: Control of steatorrhea was defined as a less than 30 percent (%) of fat in stools as measured by nuclear magnetic resonance (NMR) spectroscopy in all stool samples which are collected at baseline phase (usual pancreatic enzymes) during which the patients were on their prescribed pancreatic enzyme product (PEP) and during the 5-day collection period of the treatment phase during which the PEP was replaced with Ultrase MT12.
Time Frame: A period of 19 to 24 days, from Baseline (Visit 2) to Day 15 to19 of Treatment Phase (Visit 3)
Population: The Intent-to-treat (ITT) population included all patients who signed an informed consent form (ICF) and started the baseline phase. The 50th percentile imputation method was used for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ultrase® MT12
Number analyzed (Participants) | 49
percentage of patients
  Baseline phase (usual pancreatic enzymes) | 46.9 [32.5 to 61.7]
  Treatment phase | 42.9 [28.8 to 57.8]

2. Secondary Outcome: Percentage of Patients With Normal Stool Frequency
Description: Normal stool frequency was defined as having less than 4 bowel movements per day in baseline phase (usual pancreatic enzymes) during which the patients were on their prescribed pancreatic enzyme product (PEP) and 5-day collection period of the Treatment Phase during which the PEP was replaced with Ultrase MT12.
Time Frame: A period of 19 to 24 days, from Baseline (Visit 2) to Day 15 to19 of Treatment Phase (Visit 3)
Population: The ITT population included all patients who signed an ICF and started the baseline phase. Here "n" signifies patients who were evaluable for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ultrase® MT12
Number analyzed (Participants) | 49
percentage of patients
  Baseline phase (usual pancreatic enzymes): n=49 | 87.8 [75.2 to 95.4]
  Treatment phase: n=45 | 91.1 [78.8 to 97.5]

3. Secondary Outcome: Percentage of Stools With Normal Consistency
Description: Normal consistency of stool was defined as hard and formed or soft and formed consistency. Abnormal consistency was defined as loose and unformed stool or liquid stools and diarrhea. Percentage of stools with normal consistency of each patient was calculated from normal consistency of stools by the patient per day. Mean percentage of stools with normal consistency in baseline phase (usual pancreatic enzymes) during which the patients were on their prescribed pancreatic enzyme product (PEP) and 5-day collection period of the treatment phase during which the PEP was replaced with Ultrase MT12, for total patients was summarized.
Time Frame: A period of 19 to 24 days, from Baseline (Visit 2) to Day 15 to19 of Treatment Phase (Visit 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of stools
Arm/Group | Ultrase® MT12
Number analyzed (Participants) | 49
percentage of stools
  Baseline phase (usual pancreatic enzymes): n=49 | 77.38 (24.274)
  Treatment phase: n=45 | 76.03 (23.161)

4. Secondary Outcome: Percentage of Stools With Abnormal Characteristics
Description: Stools of abnormal characteristics were defined as bulky/large, foul-smelling and/or oily stools. Mean percentage of stools with abnormal characteristics in baseline phase (usual pancreatic enzymes) during which the patients were on their prescribed pancreatic enzyme product (PEP) and 5-day collection period of the treatment phase during which the PEP was replaced with Ultrase MT12, for total patients was summarized.
Time Frame: A period of 19 to 24 days, from Baseline (Visit 2) to Day 15 to19 of Treatment Phase (Visit 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of stools
Arm/Group | Ultrase® MT12
Number analyzed (Participants) | 49
percentage of stools
  Baseline phase (usual pancreatic enzymes): n=49 | 70.37 (30.037)
  Treatment phase: n=45 | 61.13 (33.582)

5. Secondary Outcome: Mean Number of Days Without Abdominal Complaints
Description: Abdominal complaints were defined as the reporting of abdominal pain and/or unusual and excessive flatulence/gas production. Mean number of days without abdominal complaints in baseline phase (usual pancreatic enzymes) during which the patients were on their prescribed pancreatic enzyme product (PEP) and 5-day collection period of the treatment phase during which the PEP was replaced with Ultrase MT12, for total patients was summarized.
Time Frame: A period of 19 to 24 days, from Baseline (Visit 2) to Day 15 to19 of Treatment Phase (Visit 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ultrase® MT12
Number analyzed (Participants) | 49
days
  Baseline phase (usual pancreatic enzymes): n=49 | 2.0 (1.89)
  Treatment phase: n=45 | 2.3 (2.08)

6. Other Pre Specified Outcome: Total Weight of Stools
Description: The total weight of stools in grams (g) is the total weight obtained during the stool collection period regardless of the number of stools that had been collected during this same collection period. Mean total weight of stools in baseline phase (usual pancreatic enzymes) during which the patients were on their prescribed pancreatic enzyme product (PEP) and 5-day collection period of the treatment phase during which the PEP was replaced with Ultrase MT12, for total patients was summarized.
Time Frame: A period of 19 to 24 days, from Baseline (Visit 2) to Day 15 to19 of Treatment Phase (Visit 3)
Population: The ITT population included all patients who signed an ICF and started the baseline phase. Here "N" (number of patients analyzed) represents number of patients who were evaluable for this outcome measure. Here "n" signifies patients who were evaluable for each specified category.
Measure: Mean (Standard Deviation); unit: gram (g)
Arm/Group | Ultrase® MT12
Number analyzed (Participants) | 48
gram (g)
  Baseline phase (usual pancreatic enzymes): n=48 | 349.2 (144.40)
  Treatment phase: n=45 | 367.0 (155.85)

7. Other Pre Specified Outcome: Percentage of Days With Abdominal Pain and Excessive Flatulence
Description: Mean percentage of days with abdominal complaints during baseline phase (BP) and the 5-day collection period of the treatment phase for total patients was summarized. Abdominal complaints were defined as the reporting of abdominal pain and/or unusual and excessive flatulence/gas production. Mean number of days abdominal pain (AP) and excessive flatulence (EF) in baseline phase (usual pancreatic enzymes) during which the patients were on their prescribed pancreatic enzyme product (PEP) and 5-day collection period of the treatment phase during which the PEP was replaced with Ultrase MT12, for total patients was summarized.
Time Frame: A period of 19 to 24 days, from Baseline (Visit 2) to Day 15 to19 of Treatment Phase (Visit 3)
Population: The ITT population included all patients who signed an ICF and started the baseline phase. Here "n" signifies patients who were evaluable for each specific category.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Ultrase® MT12
Number analyzed (Participants) | 49
percentage of days
  BP (usual pancreatic enzymes): AP (n=48) | 12.50 (27.250)
  Treatment phase: AP (n=44) | 9.20 (20.056)
  BP (usual pancreatic enzymes): EF (n=49) | 52.04 (37.582)
  Treatment phase: EF (n=45) | 45.56 (42.080)

8. Post Hoc Outcome: Percentage of Patients With Control of Steatorrhea Based on Concomitant Use of Proton Pump Inhibitors (PPIs)
Description: Control of steatorrhea was defined as a less than 30 percent (%) of fat in stools as measured by nuclear magnetic resonance (NMR) spectroscopy in all stool samples which are collected in baseline phase (usual pancreatic enzymes) during which the patients were on their prescribed pancreatic enzyme product (PEP) and 5-day collection period of the treatment phase during which the PEP was replaced with Ultrase MT12.
Time Frame: A period of 19 to 24 days, from Baseline (Visit 2) to Day 15 to19 of Treatment Phase (Visit 3)
Population: The ITT population included all patients who signed an ICF and started the baseline phase. There was no imputation of missing data. Here "n" signifies patients who were evaluable for each specific category.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ultrase® MT12
Number analyzed (Participants) | 49
percentage of patients
  BP (usual pancreatic enzymes): With PPIs (n=28) | 53.6 [33.9 to 72.5]
  Treatment phase: With PPIs (n=26) | 53.8 [33.4 to 73.4]
  BP (usual pancreatic enzymes): Without PPIs(n=20) | 40.0 [19.1 to 64.0]
  Treatment phase: Without PPIs (n=19) | 36.8 [16.3 to 61.6]

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to the study discharge (last study visit on Day 24 of treatment phase or early discontinuation visit)
Description: Safety population included patients who signed an ICF, completed the baseline phase and started the treatment phase by taking at least one dose of the study treatment. Adverse event (AE) was defined as any untoward medical occurrence regardless of causal relationship to study medication.
Arm/Group | Ultrase® MT12
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 24/48
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ultrase® MT12 (N=48)
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 4
Feacal fat increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions vary in accordance with each agreement with the individual investigators. Sponsor will allow publication after a multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and can defer publication for a period of time to allow for Sponsor to obtain patent or other intellectual property right protection.